CLINICAL TRIAL: NCT06925997
Title: Metabolic Effects of Endogenous Bile Acids After Gastric Bypass Surgery
Acronym: Bile-bar
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Marie-Louise Dichman, Principal investigator, MD, Ph.D. student, Hvidovre University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: H-22041713
Record Dates: First submitted 2024-04-15; First posted 2025-04-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Bariatric Surgery Candidate; Bile Acid, Elevated Serum; Glucose Metabolism Disorders
MeSH Terms: conditions — Glucose Metabolism Disorders | interventions — Colesevelam Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 3.75 mg Colesevelam in 8 weeks (Experimental)
  Interventions: Drug: Colesevelam

INTERVENTIONS:
Drug: Colesevelam — Colesevelam is an approved drug with well known adverse events. Gastrointestinal side effects (Obstipation, flatulence, abdominal pain, diarrhea, nausea, meteorism, vomiting, chanced faeces) are very common (>10%) or common (1-10%), but are mild and tolerable in most cases. All participants will be monitored closely, and colesevelam will be discontinued if the subject experience unreserved adverse events. All effects of colesevelam are transient (17-19) as the compound is not absorbed to the systemic circulation, i.e. treatment effects cease when the drug is excreted from the intestine. Specifically, no permanent metabolic effects of colesevelam has been observed in crossover experiments (27). Therefore, 8 weeks of colesevelam treatment as planned in the current study will have no long lasting positive or negative effects on the participants.

SUMMARY:
Non-randomized, open-label, parallel-group clinical study evaluating the effects of endogenous bile acids on changes in plasma fibroblast growth factor-19 (FGF-19) and glucose metabolism by extended depletion of circulating bile acids using colesevelam as an experimental tool in subjects operated with gastric by-pass (RYGB).

DETAILED DESCRIPTION:
The study design consists of 4 study visits, two performed before (V1 at day -7 and V2 at day 0 relative to initiation colesevelam treatment) and two after approximately 8 weeks of colesevelam treatment (V3 at day 49 and V4 at day 56). Biometrics, fasting blood samples and a standard mixed meal test are performed at V2 and V4. 75Se-HCAT scintigraphy is carried out between V1 to V2 and V3 to V4, respectively. Between V2 and V3 the subjects will have two telephone calls and one visit at the Endocrine Research Unit for fasting blood samples to make sure they do not experience any adverse events and are compliant.

The control groups will only participate in V1 and V2. The aim with the control groups is to have baseline values for unoperated subjects with and without diabetes to compare with the values in the intervention group after 8 weeks of depletion of endogenous bile acids.

ELIGIBILITY:
Inclusion Criteria:

Intervention group

* RYGB-operated ≥ 18 months prior to inclusion
* History of diabetes prior to RYGB (HbA1c ≥48 mmol/mol or use of antidiabetic medication)
* HbA1c <58 mmol/mol on no antidiabetic medication or metformin alone
* Weight change < ±3 kg for >3 months at time of inclusion

Control group A

* No history of diabetes
* HbA1c <48 mmol/mol at time of inclusion
* Fasting plasma glucose < 7.0 mmol/L at time of inclusion
* Weight change < ±3 kg for >3 months at time of inclusion Control group B
* Type 2 diabetes (HbA1c ≥48 mmol/mol or use of antidiabetic medication at time of inclusion)
* Weight change < ±3 kg for >3 months at time of inclusion

Exclusion Criteria:

* Pregnancy or breastfeeding
* Haemoglobin < 6.5 mmol/L at time of inclusion
* Fasting plasma glucose > 10.0 mmol/L at time of inclusion
* Prior cholecystectomy
* Chronic or tendency to diarrhoea

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-05-02 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Glucose | 8 weeks
  Changes in total areal under the curve (AUC) of plasma glucose concentrations during the mixed meal test after 8 weeks of colesevelam-induced depletion of endogenous bile acids (V4) compared with baseline in the intervention group (V2).
FGF-19 | 8 weeks
  Changes in total AUC of plasma FGF-19 concentrations during the mixed meal test after 8 weeks of colesevelam-induced depletion of endogenous bile acids (V4) compared with baseline in the intervention group (V2).

OTHER OUTCOMES:
Explorative outcomes, glucose | 8 weeks
  Plasma glucose concentration during the mixed meal test after 8 weeks of colesevelam-induced depletion of endogenous bile acids (V4) compared with baseline in the intervention group (V2).
Explorative outcomes, Bile acids | 8 weeks
  after 8 weeks of colesevelam-induced depletion of endogenous bile acids (V4) compared with baseline in the intervention group (V2).
Explorative outcomes, FGF-19 | 8 weeks
  after 8 weeks of colesevelam-induced depletion of endogenous bile acids (V4) compared with baseline in the intervention group (V2).
Explorative outcomes, cholecystokinin (CCK) | 8 weeks
  after 8 weeks of colesevelam-induced depletion of endogenous bile acids (V4) compared with baseline in the intervention group (V2).
Explorative outcomes, glucagon-like peptide-1 (GLP-1) | 8 weeks
  after 8 weeks of colesevelam-induced depletion of endogenous bile acids (V4) compared with baseline in the intervention group (V2).
Explorative outcomes, Neurotensin | 8 weeks
  after 8 weeks of colesevelam-induced depletion of endogenous bile acids (V4) compared with baseline in the intervention group (V2).
Explorative outcomes, triglycerides | 8 weeks
  after 8 weeks of colesevelam-induced depletion of endogenous bile acids (V4) compared with baseline in the intervention group (V2).
Explorative outcomes, cholesterol | 8 weeks
  after 8 weeks of colesevelam-induced depletion of endogenous bile acids (V4) compared with baseline in the intervention group (V2).
Explorative outcomes, C4 concentrations | 8 weeks
  after 8 weeks of colesevelam-induced depletion of endogenous bile acids (V4) compared with baseline in the intervention group (V2).
Explorative outcomes, insulin sensitivity | 8 weeks
  Changes in Insulin sensitivity (HOMA-IR) after 8 weeks of colesevelam-induced depletion of endogenous bile acids (V4) compared with baseline in the intervention group (V2).
Explorative outcomes, betal-cell function | 8 weeks
  Changes in Beta-cell function (disposition index) after 8 weeks of colesevelam-induced depletion of endogenous bile acids (V4) compared with baseline in the intervention group (V2).
Explorative outcomes, bile acid retention | 8 weeks
  Changes in Insulin bile acid retention (75Se-HCAT) after 8 weeks of colesevelam-induced depletion of endogenous bile acids (V4) compared with baseline in the intervention group (V2).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medicine, Copenhagen University Hospital - Amager and Hvidovre, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: Undecided